CLINICAL TRIAL: NCT06013995
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986326 in Adult Participants With Discoid Lupus Erythematosus, Subacute Cutaneous Lupus Erythematosus, or Systemic Lupus Erythematosus
Brief Title: A Study to Investigate the Safety, Tolerability, Drug Levels and Drug Effects of BMS-986326 in Adult Participants With Different Forms of Lupus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM034-1000; 2022-503009-39 (Other: EU CTR)
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Lupus
Keywords: Pharmacokinetics; BMS-986326; Cutaneous Lupus; discoid lupus erythematosus (DLE); subacute cutaneous lupus erythematosus (SCLE); Systemic lupus erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Discoid; Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A: BMS-986326 Dose 1 IV (Experimental)
  Interventions: Drug: BMS-986326; Other: Placebo for BMS-986326
- Cohort B: BMS-986326 Dose 2 IV (Experimental)
  Interventions: Drug: BMS-986326; Other: Placebo for BMS-986326
- Cohort C1: BMS-986326 Dose 3 IV (Experimental)
  Interventions: Drug: BMS-986326; Other: Placebo for BMS-986326
- Cohort C2: BMS-986326 Dose 3 SC (Experimental)
  Interventions: Drug: BMS-986326; Other: Placebo for BMS-986326
- Cohort D2: BMS-986326 Dose 4 SC (Experimental)
  Interventions: Drug: BMS-986326; Other: Placebo for BMS-986326
- Cohort E2: BMS-986326 Dose 3 SC (Experimental)
  Interventions: Drug: BMS-986326; Other: Placebo for BMS-986326

INTERVENTIONS:
Drug: BMS-986326 — Specified dose on specified days
Other: Placebo for BMS-986326 — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate safety, drug levels and drug effects on cells and organs of the body, after receiving multiple increasing doses of BMS-986326 via intravenous (IV) infusion or subcutaneous (SC) injection, in participants with different forms of lupus.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Discoid Lupus Erythematosus (DLE), Subacute Cutaneous Lupus Erythematosus (SCLE), or Systemic Lupus Erythematosus (SLE).
* Participants with DLE or SCLE must have their diagnosis at least 3 months prior to screening and must be confirmed by biopsy (except if only the facial/head/neck region is affected) and must have some ongoing disease activity (based CLASI-A scoring).
* Participants with SLE must have a diagnosis of SLE at screening based on the 2019 EULAR/ACR Classification for SLE and have mild-moderate disease severity (based on a SLEDAI-2K score).

Exclusion criteria:

* SLE that is considered by the Investigator to be severe.
* Drug-induced CLE and drug-induced SLE.
* Women who are pregnant or breastfeeding.
* Current use of >10 mg prednisone (or equivalent) per day.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 228 days
Number of participants with serious adverse events (SAEs) | Up to 228 days
Number of participants with clinical laboratory abnormalities | Up to 228 days
Number of participants with vital sign abnormalities | Up to 228 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 228 days
Number of participants with physical examination abnormalities | Up to 228 days

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Predose and post-dose up to Day 167
Time of Cmax (Tmax) | Predose and post-dose up to Day 167
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-T]) | Predose and post-dose up to Day 167
Serum PK parameters such as AUC(TAU) | Predose and post-dose up to Day 167
Change from baseline in regulatory T cells (Treg) count to Day 144 | Baseline up to Day 144
Change from baseline in Treg-to-conventional t cells (Tconv) ratio | Baseline up to Day 144
Number of participants with anti-drug antibodies | Baseline up to Day 167

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (11):
  - Local Institution - 0048, San Diego, California
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - North Georgia Rheumatology, Lawrenceville, Georgia
  - Skin Sciences, Louisville, Kentucky
  - Local Institution - 0062, Las Vegas, Nevada
  - Columbia University Irving Medical Center, New York, New York
  - Local Institution - 0005, Duncansville, Pennsylvania
  - Allen Arthritis, Allen, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
- Argentina (2):
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Clinica Adventista Belgrano, CABA, Buenos Aires F.D.
- Local Institution - 0072, Sofia, Bulgaria
- Germany (3):
  - Charité Research Organisation, Berlin
  - Städtisches Klinikum Dessau, Dessau
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
- Mexico (3):
  - Local Institution - 0073, Cuauhtémoc, Ciudad de México, DIF
  - Local Institution - 0068, Mexico City, DIF
  - Local Institution - 0077, Chihuahua City
- Local Institution - 0051, Leiden, Netherlands
- Poland (2):
  - Local Institution - 0074, Poznan
  - Local Institution - 0069, Warsaw
- Romania (2):
  - Local Institution - 0065, Bucharest, București
  - Local Institution - 0064, Cluj-Napoca, Cluj
- Spain (2):
  - Local Institution - 0046, A Coruña, A Coruña [La Coruña]
  - Local Institution - 0045, Córdoba, Córdoba

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06013995.html